CLINICAL TRIAL: NCT02228213
Title: A Phase 2B Randomised, Double-Blind, Placebo-Controlled Trial of the Efficacy and Safety of MIS416 in the Treatment of Subjects With Secondary Progressive Multiple Sclerosis
Brief Title: Safety and Efficacy Study of MIS416 to Treat Secondary Progressive Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Innate Immunotherapeutics (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIS416-202; U1111-1166-0910 (Other: WHO)
Record Dates: First submitted 2014-08-21; First posted 2014-08-28 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Secondary Progressive Multiple Sclerosis
Keywords: multiple sclerosis; SPMS
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — MIS416 vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): 500 mcg MIS416 500 at 0.2 mg/mL administered i.v. once weekly for 52 weeks
  Interventions: Biological: MIS416
- Saline (Placebo Comparator): Saline administered i.v. once weekly for 52 weeks
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: MIS416 — Intravenous administration weekly for 52 weeks
  Arms: Treatment
Drug: Saline — Intravenous administration weekly for 52 weeks
  Other Names: Placebo
  Arms: Saline

SUMMARY:
The purpose of this study is to determine whether MIS416 administered once weekly over 12 months is safe, tolerable, and improves a range of signs and symptoms associated with secondary progressive multiple sclerosis.

DETAILED DESCRIPTION:
The primary objectives of the study are to:

1. Determine the efficacy of MIS416, relative to placebo, when administered repeatedly via weekly intravenous (IV) administration to subjects with Secondary Progressive Multiple Sclerosis, as assessed by its effect on measures of neuromuscular function.
2. Determine the safety and tolerability of a weekly regimen of MIS416.

The secondary objectives of the study are to:

1. Determine the effect of MIS416 on disease activity and neurodegeneration by assessing changes in Magnetic Resonance Imaging (MRI) markers including lesions, whole brain atrophy (WBA) and Magnetization Transfer Ratio (MTR).
2. Determine the effect of MIS416 on Patient Reported Outcomes (PRO) related to disability and health status.
3. Assess, in a subset of subjects, the pharmacodynamic (PD) effects of MIS416, including effects on serum, Peripheral Blood Mononuclear Cell (PBMC), and Cerebral Spinal Fluid (CSF) cytokine/chemokine levels and expression patterns.

ELIGIBILITY:
Inclusion Criteria:

1. A historical or current cranial MRI scan demonstrating T2-hyperintense lesions consistent with MS.
2. Has SPMS as determined by the 2010 Update to the McDonald Criteria
3. An Expanded Disability Status Scale (EDSS) of 3.0 to 6.5 at Screening.
4. Has SPMS which, in the judgment of the investigator, has been clinically active and functionally progressive within the 2 years prior to Screening
5. The absence of MS relapse for at least two years prior to Baseline.
6. Neurologically stable for at least four weeks prior to Screening.
7. Has the following laboratory values within three days prior to initiation of Investigational Product:

   * Absolute neutrophil count (ANC) >= 1 x 109/L;
   * Platelet count >= 100 x 109/L;
   * Serum creatinine =< 1.5 mg/dL;
   * Aspartate aminotransferase (AST) =<2 × upper limit of normal;
   * Alanine aminotransferase (ALT) =< 2 × upper limit of normal.
8. Provided written informed consent to participate.

Exclusion Criteria:

1. Has primary Progressive MS (PPMS), Relapsing Remitting (RRMS), or progressive relapsing MS as determined by the 2010 update to the McDonald Criteria.
2. Has not completed the discontinuation period for approved and/or investigational multiple sclerosis disease modifying therapies prior to screening.
3. Has had any other immunomodulatory drug therapy or immunosuppressive therapy within four weeks prior to Screening, or systemic corticosteroids within the eight weeks prior to Screening.
4. Any previous exposure to investigational MS therapeutic vaccines.
5. Any use of cell-depleting monoclonal antibodies including, but not limited to, Rituximab, or Ocrelizumab.
6. A diagnosis or history of collagen vascular disease (including Sjögren's syndrome and systemic lupus erythematosus), anticardiolipin antibody syndrome, cerebral autosomal dominant arteriopathy with subcortical infarcts and leukoencephalopathy, sarcoidosis, vasculitis, Behcet's syndrome and/or Lyme disease.
7. Contraindication to MRI (e.g., pacemaker or other contraindicated implanted metal device, allergy to gadolinium, or unmanageable claustrophobia).
8. A history of alcohol or drug abuse (including cannabinoid use) within two years prior to Screening.
9. Has had major surgery or radiation therapy within four weeks prior to Screening.
10. Has an active infection requiring antibiotics within two weeks prior to Screening.
11. Has had active malignancy within two years of Screening, with the exception of basal cell carcinoma and squamous cell carcinoma of the skin.
12. Uncontrolled congestive heart failure, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, or transient ischemic attack within twelve weeks prior to Screening.
13. Has angina, other symptomatic coronary artery disease, or known cardiomyopathy.
14. Has symptomatic cardiac dysrhythmias requiring treatment, or persistent prolongation of the QTcF (Fredericia) interval to > 450 msec for males or > 470 msec for females.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2014-10; Primary Completion 2017-05 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of neuromuscular function at 12 months | Baseline, 3, 6, 9 and 12 months
  Neuromuscular function will be assessed using the following test:
  * MS Function Composite (MSFC), comprising the; timed 25 Foot Walk, 9 Hole Peg Test (9HPT), and Paced Auditory Serial Addition Test (PASAT);
  * Jebsen Hand Function Test (JHFT);
  * Grip, tip and key pinch strength;
  * Symbol digit modalities test (SDMT);
  * Sloan low-contrast letter visual acuity (SLCVA);
  * 6-minute walk test (6MWT);
Proportion of Participants with Serious and Non-Serious Adverse Events | Up to 12 months
  Safety assessments will be conducted at each study visit and include; characterization of the type, incidence, severity, timing, seriousness, and relationship to treatment of adverse events (AEs); effects on vital signs and clinical laboratory parameters; changes on electrocardiograms (ECGs); and at 3 months and 12 months - the number of gadolinium-enhancing lesions on cranial MRI assessments.

SECONDARY OUTCOMES:
Change from baseline of disability and health status at 12 months | Baseline, 3, 6, 9, and 12 months
  Disability and health status will be assessed using the following assessments and patient reported outcomes:
  * Expanded Disability Status Scale (EDSS)
  * Patient Reported Outcomes (PROs) including;
    * SF-36 and its components;
    * MS Impact Scale (MSIS-29);
    * Neurological Fatigue Index for MS (NFI-MS);
    * Brief Pain Inventory (BPI).
Change from baseline of neurodegeneration by assessing changes in Magnetic Resonance Imaging (MRI) markers at 12 months | Baseline, 3, and 12 months
  Disease activity and neurodegeneration will be assessing using Magnetic Resonance Imaging (MRI) markers including lesions, whole brain atrophy (WBA) and Magnetization Transfer Ratio (MTR).
Change from baseline of activity of immune biomarkers in serum | Up to 1 year
  The effect on immune biomarkers will include the analysis of serum for some or all of the following markers: IP-10 (CXCL10), MCP-1 (CCL2), MIG (CXCL9), IL-8 (CXCL8), IFNγ, Neopterin, IL-1RA, sTNF-R, IL-12/23, p40, CD62E (E-selectin), CD54 (ICAM-1), and CD106 (VCAM-1).
Change from baseline of activity of immune biomarkers in cerebrospinal fluid (CSF) | Up to 12 months
  The effect on immune biomarkers will include the analysis of CSF for some or all of the following markers: IP-10 (CXCL10), MCP-1 (CCL2), MIG (CXCL9), IL-8 (CXCL8), IFNγ, Neopterin, IL-1RA, sTNF-R, IL-12/23, p40, CD62E (E-selectin), CD54 (ICAM-1), and CD106 (VCAM-1).
Change from baseline in Peripheral Blood Mononuclear Cell (PBMC) immune biomarkers | Up to 12 months
  Some or all of these biomarkers may be assayed ex vivo: PBMC expression of mRNA encoding proteins involved in myeloid differentiation and immune regulatory function (e.g. VEGF, Arginine, INOS, IL-10, MMP9); PBMC myeloid subset production of IL-10, TGFβ, IL-6, TNFα, IL-1β, IFNγ, IL-17, and GM-CSF in response to stimulation with LPS, LPS/IFNγ or MIS416 ex vivo; and PBMC subset analysis of myeloid and dendritic cell subsets for immunoregulatory cell subset markers.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, Study Director — Innate Immunotherapeutics
Locations (7):
- Australia (5):
  - The Wesley-St. Andrew's Research Institute, Brisbane, Queensland
  - PARC Clinical Research, Adelaide, South Australia
  - Nucleus Network - Centre for Clinical Studies, Melbourne, Victoria
  - Western Australian Neuroscience Research Institute, Perth, Western Australia
  - Neurodegenerative Disorders Research, West Perth, Western Australia
- New Zealand (2):
  - Optimal Clinical Trials, Auckland
  - P3 Research, Wellington